CLINICAL TRIAL: NCT05071339
Title: GnRH Antagonist Pre-treatment in the Early Follicular Phase for the Prevention of Asynchronous Follicular Growth - A Proof-of-concept Pilot Study
Brief Title: GnRH Antagonist Pre-treatment for the Prevention of Asynchronous Follicular Growth
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Assaf Harofeh MC, Senior physician, Assaf-Harofeh Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0013-21-ASF
Record Dates: First submitted 2021-02-20; First posted 2021-10-08 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: IVF
MeSH Terms: interventions — ganirelix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Participants (Experimental): Patients treated at the IVF unit at Shamir Medical Center planned for an antagonist cycle will undergo blood test and US exam at day 2-3 of their menstrual cycle. Patients will be recruited if a leading follicle 10-13 is shown in the presence of E2 > 200-350 pmol/L.
  Patients will start GnRH antagonist injections [Cetrotide (cetrolix) or Orgalutran (ganirelix) - depending on their primary prescription] for 3-5 days intervention.
  Interventions: Drug: Ganirelix Acetate, Cetrolix Acetate

INTERVENTIONS:
Drug: Ganirelix Acetate, Cetrolix Acetate — 3-6 days of 0.25mg GnRH antagonist starting day 2-3 of the menstrual cycle prior to the administration of the original protocol.

SUMMARY:
In the study the investigators would like to examine the effect of GnRH antagonist administration at the beginning of the follicular phase in patients presenting with high baseline estradiol levels of 200 pmol/L or above with a leading follicle of 11-13 mm. In the unit's practice, patients presenting for cycle initiation with a leading follicle > 10 in the presence of E2 > 200 pmol/L (54 pg/ml) are deferred and receive a priming antagonist protocol in their sequential cycle. The aim of this intervention is to suppress FSH levels at the beginning of the cycle thus preventing estradiol secretion of the leading follicle. This may contribute to better synchronization of the remaining antral follicles cohort and allow for a better cycle outcome instead of cancellation or one-month postponement. As previous studies using GnRH antagonist pre-treatment prior to GT initiation for synchronization purposes demonstrated positive results (including different patient population) , no deleterious effects are expected.

DETAILED DESCRIPTION:
During the late luteal phase, parallel to the corpus luteum demise, FSH levels gradually increase in order to preserve antral follicles from atresia. Early antral follicles show different sensitivity to FSH possibly contributing to the establishment of the dominant follicle by starting their development earlier than others. Previous studies indicated larger follicles are more sensitive to FSH then smaller ones, thus respond to lower levels of FSH. The premature gradual exposure to FSH may accelerate the development of the larger follicle and accentuate size discrepancies observed during controlled ovarian hyperstimulation (COH).

During COH exogenous gonadotropins are expected to influence early antral follicle growth to simultaneously reach functional and morphological maturation. Significant size discrepancy at the time of HCG administration may result in a larger fraction of immature oocytes, reducing the number of embryos and the pregnancy rate.

Since baseline FSH levels are higher in older and poor responder patients, early antral follicles are exposed to higher levels of FSH thus size discrepancies are observed more frequently, contributing to higher cancellation rates and reducing furthermore pregnancy rates.

Several protocols have been established to overcome early antral follicle exposure to FSH. Estradiol priming for 7 days in the late luteal phase prior to GT stimulation achieved FSH suppression and resulted in size discrepancy reduction and better cycle outcome (higher number of mature oocytes, embryos and pregnancy rates). A meta-analysis demonstrated reduced cycle cancellation rate and higher clinical pregnancy rate. GnRH antagonist priming, also by reducing FSH levels in the late luteal phase, resulted in coordination of early antral follicular size. These priming protocols require preplanning and a relatively predictable menstrual cycle in order to start the priming supply in the late luteal phase. Poor responder patients and those in-between IVF treatment cycles may not have regular menses or may be waiting for pregnancy test results, thus do not represent optimal potential candidates for a priming protocol.

Several studies have investigated the outcome of GnRH antagonist supplementation at the beginning of the menstrual cycle prior to GT stimulation. The delayed start protocol which combines estradiol priming followed by GnRH antagonist for 7 days at the beginning of menses prior to GT administration to further synchronize antral follicles improved ovarian response in poor responders and reduced cycle cancellation rate with no significant effect on pregnancy rates. A preliminary study investigated the effect of three day administration of GnRH antagonist at the beginning of the follicular phase prior to GT stimulation in normal responders regardless of baseline hormonal levels and found a trend towards increase in clinical pregnancy rate, and similar profiles of early embryo development, compared to standard fixed GnRH antagonist protocol.

Patients not receiving priming protocol that are planned for an antagonist protocol usually start their stimulation on day 2-3 of menses. A baseline Ultrasound and hormonal blood test are performed to determine adequacy of cycle start. In a long agonist protocol, gonadotropin stimulation begins after confirming that effective pituitary downregulation has been achieved (serum estradiol level <30-40 pg/mL, no follicles >10 mm in diameter). In an antagonist protocol cut offs may be defined according to the clinical observations and expectations of each individual program. There have been reports of estradiol level cut-offs between 56pg/ml and 80pg/ml with an average of 35pg/ml. In a prospective randomised trial Patients who presented with an elevated day 3 E2 >80 pg/mL in a cycle before IVF-ET had a higher cancellation rate and achieved a lower PR independent of FSH level.

In summary, several studies have proposed the use of different priming modalities in order to suppress the early rise of FSH at the late luteal stage, including the use of estrogen and GnRH-antagonist. No study examined the effect of these modalities on women with follicular and hormonal levels suggesting early recruitment and beginning of development of the leading follicle.

Study aim: In this study the investigators would like to examine the effect of GnRH antagonist administration at the beginning of the follicular phase in patients presenting with high baseline estradiol levels of 200 pmol/L or above (<350) with a leading follicle of 10-13 mm. In the unit's practice, patients presenting for cycle initiation with a leading follicle > 10 in the presence of E2 > 200 pmol/L (54 pg/ml) are deferred and receive a priming antagonist protocol in their sequential cycle. The aim of this intervention is to suppress FSH levels at the beginning of the cycle thus preventing estradiol secretion of the leading follicle. This may contribute to better synchronization of the remaining antral follicles cohort and allow for a better cycle outcome instead of cancellation or one-month postponement. As previous studies using GnRH antagonist pre-treatment prior to GT initiation for synchronization purposes demonstrated positive results (including different patient population) , no deleterious effects are expected.

Materials and Methods: This is a proof-of-concept pilot study. Patients will be recruited at the reproductive medicine unit of Shamir Medical Center, Israel.

Study population: Patients undergoing controlled ovarian hyper stimulation at the IVF unit, Shamir medical center. Planned recruitment of 15 patients.

Sample size: This is a proof of concept pilot study to evaluate the feasibility and potential effectiveness of the intervention. A sample size of 15 patients will allow detecting the potential for use of cycles that would have been cancelled using standard protocols. As the comparator is mandatory cancellation, i.e. 0% use of cycles, this sample size is sufficient.

Study protocol:

Patients treated at the IVF unit at Shamir Medical Center planned for an antagonist cycle will undergo blood test and US exam at day 2-3 of their menstrual cycle. Patients will be recruited if a leading follicle > 10mm is shown in the presence of E2 200-350pmol/L. Following the initial US exam in the morning, if a follicle 10-13 mm will be demonstrated, the patient will receive a form explaining that the protocol may be changed according to blood test results with three possible options: 1. Continuation with the original protocol 2. Cancellation 3. Change in protocol as part of a research if the patient agrees to participate. As patients undergo blood draws in the morning, with results available in the afternoon, the initial recruitment will be performed over the phone with signed informed consent received at the following clinic visit.

Patients will receive a verbal explanation over the phone and following verbal consent will start GnRH antagonist injections [Cetrotide (cetrolix) or Orgalutran (ganirelix) - depending on their primary prescription] for 3-5 days by which time a second blood test (for estradiol, progesterone, LH and FSH) and US exam will be performed.

* If estradiol levels have decreased to < 200 pmol/L then ovarian stimulation according to the original patient's protocol will be started.
* If estradiol levels have increased above 5%, the cycle will be cancelled.
* If estradiol levels have slightly decreased but still above 200 or increased in less than 5% then GnRH antagonist for 3 more days will be prescribed. After these 3 days if estradiol levels have decreased to < 200, ovarian stimulation according to the original patient's protocol will be started. If estradiol levels are > 200 then cycle will be cancelled.

When treatment is continued, the previous leading follicle will be separately followed. Treatment outcomes will be recorded, including the number of large and small follicles, number of mature oocytes of expected mature oocytes and number of embryos. Leading follicle outcome will be recorded separately. In patients with a previous or a subsequent cycle with similar GT dosages, cycle outcomes will be compared to the cycle with the intervention.

Risks to subjects: No anticipated risks over regular stimulation protocol side effects.

Statistical analyses: Descriptive statistics will be used.

ELIGIBILITY:
Inclusion Criteria:

* Planed antagonist protocol.
* Presentation for cycle initiation with a leading follicle 10-13 in the presence of E2 > 200 and <350 pmol/L (54 pg/ml).

Exclusion Criteria:

* Inability to provide informed consent.
* Oocyte donor

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Synchronization of follicles | 2 year
  Ratio of number of large (>15 mm) to small (<10-15mm) follicles.

SECONDARY OUTCOMES:
Number of mature oocytes that originate from the leading follicles | 2 year
  the absolute number of mature oocytes
Ratio of mature oocytes out of number of follicles | 2 year
  Number of actual oocyte yield (mature oocytes) out of expected yield (number of large follicles).
Number of oocytes compared to a previous cycle | 2 years
  Number of oocytes in the current cycle compared to the number of oocytes in a previous or future cycle using a different protocol

CONTACTS AND LOCATIONS:
Locations (1):
- Shamir Medical center, Be’er Ya‘aqov, Israel

IPD SHARING:
Plan to Share IPD: No